CLINICAL TRIAL: NCT03897660
Title: Pharmacokinetics of Omega-3 Fatty Acids Esterified in Monoglycerides, Ethyl Esters, or Triglycerides in Humans
Brief Title: MaxSimil and Vitamin K2: Determining Their Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Samuel Fortin, SFC pharma and associate professor UQAR (Unknown)
Responsible Party: Principal Investigator, Mélanie Plourde, Associate professor, Department of medicine, Geriatric service, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MaxSimil and vitamin K2
Record Dates: First submitted 2019-02-27; First posted 2019-04-01 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Omega-3 fatty acids; Vitamin K2; Bioavailability; Side effects; Monoacylglyderols
MeSH Terms: interventions — Docosahexaenoic Acids; Vitamin K 2

STUDY DESIGN:
Intervention Model Description: Double-blind controlled-randomized pharmacokinetic (PK) pilot study with crossover design (10 men and 10 women), with a minimum of 6 days between treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the research nurse will know the administration order of the different treatments administered. All plasma samples collected during the research project will be anonymized i.e. it will not be possible to identify the participant by his name since a number will be assigned to him. The code key linking the participant's name to his number will be stored, with access restricted to those designated by the principal investigator. The data file is also protected by a password.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TG form of omega-3 (Active Comparator): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive the omega-3 fatty acidsesterified in a reconstitute triglyceride form as a unique dose of 1.5 g EPA + DHA in TG form + 45 mg vitamin K2.The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: Omega-3 + vitamin K2 (TG form of omega-3)
- EE form of omega-3 (Active Comparator): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive the omega-3 fatty acids in ethyl esters form as a unique dose of 1.5 g EPA + DHA in TG form + 45 mg vitamin K2.The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: Omega-3 + vitamin K2 (EE form of omega-3)
- MaxSimil (MAG form of omega-3) (Experimental): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive the omega-3 fatty acids in MaxSimil® form as a unique dose of 1.5 g EPA + DHA in TG form + 45 mg vitamin K2.The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: Omega-3 + vitamin K2 [MaxSimil (MAG form of omega-3)]

INTERVENTIONS:
Dietary Supplement: Omega-3 + vitamin K2 (TG form of omega-3) — The intervention is a randomized double bond cross over design testing the pharmacokinetics of a monoglyceride formulation compared to a triglyceride and an ethyl ester form.
  Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours. Each participant will perform all three treatments, with a minimum of 6 days between treatments. A questionnaire will document the side effects felt by participants during the omega-3 supplement taking day.
  Arms: TG form of omega-3
Dietary Supplement: Omega-3 + vitamin K2 (EE form of omega-3) — The intervention is a randomized double bond cross over design testing the pharmacokinetics of a monoglyceride formulation compared to a triglyceride and an ethyl ester form.
  Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours. Each participant will perform all three treatments, with a minimum of 6 days between treatments. A questionnaire will document the side effects felt by participants during the omega-3 supplement taking day.
  Arms: EE form of omega-3
Dietary Supplement: Omega-3 + vitamin K2 [MaxSimil (MAG form of omega-3)] — The intervention is a randomized double blind cross over design testing the pharmacokinetics of a monoglyceride formulation compared to a triglyceride and an ethyl ester form.
  Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours. Each participant will perform all three treatments, with a minimum of 6 days between treatments. At each blood draw time points, a questionnaire will be administered to the particpant to monitor if they experiencec side effects with the dietary supplement they ingested in the morning.
  Arms: MaxSimil (MAG form of omega-3)

SUMMARY:
The benefits of a diet enriched with omega-3 fatty acids are multiple and confirmed by several clinical studies. Supplementation with vitamin K, a fat-soluble vitamin, can increase or maintain bone density in postmenopausal women and reduce the risk of fracture. In addition, some studies show that vitamin K may promote the absorption of omega-3 fatty acids. Fish oil, rich in omega-3, is one of the world's favorite forms of omega-3 supplements. However, many people suffer from gastrointestinal discomfort when ingesting fish oil capsules. To minimize these discomforts and improve plasmatic omega-3 bioavailability, Neptune Wellness Solutions has developed a patented formulation of fish oil called MaxSimil®, where omega-3s are in the monoglyceride (MAG) form, a predigested omega-3 form. This formulation has been tested in humans in a double-blind controlled-randomized pharmacokinetic (PK) pilot study with crossover design. PK is defined as a monitoring of omega-3 levels in the blood by frequent blood sampling over a period of 24 hours following the ingestion of a single dose of omega-3. The results obtained showed that MaxSimil® omega-3s are 3 times more absorbed in the blood than the comparison formulation, a source of omega-3 in the ethyl ester (EE) form.

Although this first study confirms a greater bioavailability of MaxSimil®, a complementary PK study is necessary to confirm these results and to correct an important methodological bias. In fact, the pilot study did not include a comparator group where omega-3s were in the triglyceride (TG) form, the most widely omega-3 form currently consumed, but rather use an EE form, which have lower bioavailability than TG form. This may therefore have biased the study from the point of view of the comparator and thus give the impression that the comparator had been deliberately chosen to be less bioavailable than the MaxSimil®.

In order to confirm the superiority of MaxSimil® (omega-3 MAG form), both in terms of bioavailability and incidence of side effects, the aim of this study is to redo a PK study using this time two comparators, the two main forms of omega-3 currently used (TG and EE forms), as well as a supplementation with vitamin K2 (a form of vitamin K). Our hypothesis is that MaxSimil® will be associated with a better omega-3 bioavailability and a lower incidence of side effects than the other two forms (TG and EE), and possibly also with a better vitamin K bioavailability.

DETAILED DESCRIPTION:
Long Chain-Polyunsaturated fatty acids (LC-PUFA) are needed to support normal physiological functions: Unlike saturated and monounsaturated fatty acids, synthesis of eicosapentaenoic acid (EPA, 20:5 omega-3) and docosahexaenoic acid (DHA, 22:6 omega-3) from its omega-3 PUFA precursor, alpha-linolenic acid (18:3 omega-3), is extremely limited in humans. Thus, it is recommended that DHA be obtained from dietary sources such as fish and seafood. Intake of EPA and DHA from fish normally correlates positively with the concentrations of EPA and DHA in plasma. However, recent data suggest that EPA levels are approximately twice higher in plasma lipids of the elderly as compared to young individuals, suggesting that potential alterations in EPA incorporation and utilization occur during aging. Similar results were obtained with a DHA-enriched supplement where the increase of DHA in plasma total lipids was 42% higher in the elderly compared to the young. At sufficient levels of cellular content, the LC-PUFA influence the physical nature of cell membranes and membrane protein-mediated responses, lipid-mediator generation, cell signalling, and gene expression in many different cell types. Through these mechanisms, ARA (arachidonic acid, 20:4 omega-6) and DHA influence both cell and tissue responses to external signals, and thereby their physiology. Therefore, imbalances in LC-PUFA homeostasis potentially induce dysfunctions in the physiology of organs.

Aging of the Canadians and their nutrition: Canada's population is expected to age more rapidly in the coming years. Senior citizens have become more numerous than children in 2015. A major concern about old age, both the individual and society, is a decline in health, especially if this means a loss of self-sufficiency and independence. Increasing research for promoting healthy aging is ongoing but there are physiological modifications occurring during aging that might change bioavailability of LC-PUFA. For instance, intake of EPA and DHA concentrated in fish normally correlates positively with the concentrations of EPA and DHA in plasma. However, recent data from our laboratories suggest that EPA levels are approximately twice higher in plasma lipids of the elderly as compared to young individuals, suggesting that potential alterations in EPA incorporation and utilization occur during aging. DHA response to a DHA-rich supplement was significantly higher in the elderly as compared to the young. While on DHA-rich supplement, ARA was not decreased in the young and the elderly, but similarly to EPA, ARA remained significantly higher in the elderly compared to the young. The investigators also have publish data suggesting that 40 years old is the age where the EPA and DHA levels in the plasma are higher than expected, and this was independent to their dietary omega-3 fatty acid intake. Hence, these results are important indications that the metabolism of LC-PUFA is modified by age and this observation lead to the idea that their uptake and usage by organs and tissue can be compromised.

13C-DHA in humans: Tracing metabolism of carbon 13 (13C)-labelled fatty acids may provide some insight into possible aging-related changes in fatty acid metabolism in humans. The investigators recently used 13C-DHA to trace its metabolism in six young and six elderly participants. The investigators found that, in the elderly, 13C-DHA was 4 times higher in plasma triglycerides and free fatty acids at 4 h post-dose, beta-oxidation was 1.9 times higher whereas apparent retro-conversion of 13C-DHA to other 13C-omega-3 fatty acids was 2.1 times higher 24 h and 7 d after tracer intake compared to the young. Hence, because DHA seems to remain transiently for longer periods of time in the blood of the elderly compared to the young, it may thus indicate that efficiency to remove DHA from the blood is lower in the elderly than in the young, resulting in lower incorporation of DHA in the membrane of cells that serve to initiate signalization. This observation is potentially at the root of altered signalization in the elderly compared to the young.

Bioavailability of EPA and DHA esterified in TG, PL or as an ethyl ester (EE): Most of fish oil supplements on the market are EPA and DHA esterified in TG and to a lower level in EE and PL. There has been a lot of study evaluating whether one form of esterification enhances bioavailability of EPA and DHA. In pharmacology, "Bioavailability" is defined as a subcategory of absorption and it is the portion of the administered dose of a drug or in this case, EPA+DHA that reaches the systemic circulation. By definition, an intravenous drug is 100% bioavailable but when a drug is administered orally, its bioavailability is usually decreased due to incomplete absorption or first-pass metabolism. Hence, in the review paper of Ghasemifard et al., they reviewed 21 papers that evaluated whether omega-3 fatty acid were more bioavailable when given in the form of EE, TG, non-esterified form or as a PL. Four studies were rejected because there were no control group, eight studies were evaluating pharmacokinetics (PK) defined as a follow up between 8 h up to 72 h of a single oral dose of the omega-3 fatty acid product whereas nine studies evaluated the long term intake (pharmacodynamic, PD) of a repeated daily dose of omega-3 fatty acids over a period of 2 weeks and up to 6 months. Although the methodologies of the studies differ, some conclusion about the PK was that bioavailability of EPA+ DHA was higher when given in the forms of non-esterified fatty acid > TG >>> EE. Lower absorption of the EE form might be because pancreatic hydrolysis of EPA and DHA of the EE form compared to the TG form is 10-50 times lower. Hence, the esterification form of omega-3 fatty acids might change their short-term bioavailability and this information is particularly relevant in the context of metabolic diseases that can either affect fat absorption or to an aging population where there are dyslipidemias that might change omega-3 fatty acid bioavailability.

Is MAG-Omega-3 form a better bioavailable source of EPA+DHA?: One study in rats reported bioavailability of DHA esterified in TG, PL or MAG (2-mono-acylglycerol) in plasma, erythrocytes, retina and brain tissue. They reported that after giving DHA in the different forms to rats for 35 days, DHA given in the MAG and PL form were 23-50% more concentrated in plasma total lipids and erythrocytes compared to TG-DHA. In the retina and the brain, DHA increase to the same levels whatsoever esterification form it was provided.

In conditions of lipid malabsorption, MAG enriched with EPA + DHA enhance their delivery to circulatory system in humans. In humans with cystic fibrosis, a disease recognized as having fat malabsorption, especially the long chain fatty acids such as DHA, it was reported that providing a MAG-DHA supplementation for one month was efficient to increase levels of DHA in the erythrocytes. This pilot study indicates that MAG-DHA supplementation corrects erythrocyte ARA/DHA imbalance and may exert anti-inflammatory properties. However, whether MAG-DHA is more efficient in participants without malabsorption problems remains to be established.

Side effects associated to fish oil intake: In a meta-analysis evaluating the safety and tolerability of prescribed omega-3 fatty acid supplements, it was reported that only three minor side effects were associated to fish oil intake: fishy taste, fishy burp and nausea. Although these sides effects seem limited to gastro-intestinal discomforts, it can largely compromise short- and long-term adherence to fish oil intake. One protective microorganism to gastroesophageal reflux is the presence of Helicobacter Pylori (H. Pylori). Moreover, it was recently suggested that omega-3 fatty acid supplementation inhibit H. Pylori, by inhibiting the synthesis of vitamin K that is required by this microorganism for its own survival. A pre-digested form of omega-3 fatty acid such as a MAG form with added vitamin K might limit these gastro-intestinal discomforts, and this is something the investigators want to investigate in this research project.

What is Vitamin K2?: Vitamins are essential for different physiological functions of the body. Vitamin K is a fat-soluble vitamin. Its discovery was mainly driven by its role on blood coagulation but other roles of this vitamin include regulation of calcium metabolism in tissues, cell growth and proliferation. There are three main forms for vitamin K: K1, K2 and K3. Vitamin K2 is referred as menaquinone since it shares a naphthoquinone ring and a side chain with variable length. Most of menaquinones are synthesized by bacteria. Since omega-3 fatty acid intake seems to inhibit vitamin K2 synthesis by bacteria such as H. Pylori, the investigators decided to add vitamin K2 in the MAG-omega-3 formulation to evaluate whether this formulation could decrease side effects of fish oil supplement consumption.

Rationale of this study: Over the 20th century, consumption of linoleic acid (18:2 n-6) increased from 2.79% to 7.21% of energy and this is largely due to our dependence on new food production methodologies, including soybean oil. This has created over decades a diet that is deficient in long chain omega-3 fatty acids. Recently, and because of the enthusiasm around consumption of fish oil, there is increasing concerns about fish sustainability. These critical issues leads us to have a sustainable source of omega-3 fatty acids, that is the most bioavailable and to recommend lower doses of EPA+DHA to be consumed by the population to have similar health effects. At the same time, having a source of omega-3 fatty acid with limited side effects would also contribute to a better adherence of the population to their consumption and perhaps decrease capsule waste. The plasma DHA pool is critical to bring DHA to the brain and other organs and it is dynamic, constantly exchanging FA with organs and tissues. Numerous studies have assessed the absorption, bioavailability and accretion of DHA in the plasma with the conclusion that non-esterified DHA > TG >>> EE. Recently, there has been enthusiasm for MAG-Omega-3 formulations since it was shown to improve EPA and DHA bioavailability in humans with lower intestinal lipid absorption. However, whether EPA and DHA are better absorbed and bioavailable in humans without any issues with intestinal lipid absorption remain to be established. Therefore, this project will test a MAG-Omega-3 formulation enriched with vitamin K2, since the investigators hypothesized that this formulation will be the most absorbed and bioavailable with the lowest side effects in men and women without any disease such as intestinal lipid absorption issues.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years (inclusive)
* Body mass index between 18.5 and 29.9 kg / m² (inclusive) at the pre-selection visit
* Normal to moderately elevated lipidemia (total cholesterol ≤ 240 mg / dl, LDL ≤ 160 mg / dl, TG ≤ 199 mg / dl)
* Women of childbearing potential should use an approved method of contraception for the duration of the study so that they do not become pregnant during the study

Exclusion Criteria:

* Menopause or pre-menopause with amenorrhea> 6 months
* Tobacco
* Malnutrition (assessed by albumin, hemoglobin and blood lipid levels)
* DHA plasma levels greater than 3% or people consuming omega-3 fatty acid supplements for more than one month
* History of current or past alcohol and / or drug abuse
* Parkinson's disease
* Down syndrome
* Cardiac event or recent major surgery (6 months)
* Current or past performance athlete
* Systemic disease: vasculitis, Systemic Lupus Erythematosus (SLE), sarcoidosis, cancer (unless in remission for more than 5 years and without cerebral involvement), uncompensated hypothyroidism (unless stabilized on treatment for more than 3 months), vitamin deficiency B12 not supplemented and / or complicated (unless stabilized on treatment for more than 3 months), diabetes, severe renal insufficiency
* Abnormal blood pressure and / or liver, renal or thyroid function; these conditions will not exclude a patient if he has been stabilized on treatment for at least 3 months and there has been no recent change in the medication.
* Known psychiatric history: schizophrenia, psychotic disorders, major affective disorders (bipolar disorder and major depression <5 years), panic disorder, Obsessive Compulsive Disorder (OCD)
* Epilepsy, cerebral trauma with loss of consciousness, subarachnoid hemorrhage
* Not available to perform the 3 different treatments
* Medication affecting fat absorption (i.e., Orlistat, Alli, etc.), which interferes with omega-3 fatty acids uptake (i.e., anticoagulants) or which affects lipid metabolism (i.e., all types of drug for decrease cholesterol or triglycerides)
* Nobody under a special diet like a fat-free, vegetarian or vegan diet
* People who have a malabsorption disease such as pancreatitis, Crohn's disease or who have had bariatric surgery.
* Allergy to fish or seafood
* Pregnant women or nursing women
* Person who donated blood or had significant blood loss in the 30 days prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Determine the bioavailability of omega-3 and vitamin K2 according to the forms ethyl ester (EE), triglycerides (TG) and MaxSimil® (monoglycerides, MAG): Calculating the area under the curve (AUC) 0-24h as the first parameter of the PK | Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. GC and HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours post-treatment.
  Plasma omega-3 (DHA and EPA) levels will be measured by gas phase chromatography while plasma vitamin K2 level will be measured by high-performance liquid chromatography (HPLC), each being performed randomly blindly. After GC and HPLC analyzes, area under the curve (AUC) 0-24 hours will be calculated, as the first parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of omega-3 and vitamin K2 according to the forms ethyl ester (EE), triglycerides (TG) and MaxSimil® (monoglycerides, MAG): Calculating the AUC 0-6h (absorption study) as the second parameter of the PK | Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. GC and HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours post-treatment.
  Plasma Omega-3 (DHA and EPA) will be measured by gas phase chromatography while plasma vitamin K2 will be measured by high-performance liquid chromatography (HPLC), each being performed randomly blindly. After GC and HPLC analyzes, AUC 0-6 hours (absorption study) will be calculated, as the second parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of omega-3 and vitamin K2 according to the forms ethyl ester (EE), triglycerides (TG) and MaxSimil® (monoglycerides, MAG): Calculating the maximum concentration as the third parameter of the PK | Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. GC and HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours post-treatment.
  Plasma Omega-3 (DHA and EPA) will be measured by gas phase chromatography while plasma vitamin K2 will be measured by high-performance liquid chromatography (HPLC), each being performed randomly blindly. After GC and HPLC analyzes, maximum concentration will be calculated, as the third parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of omega-3 and vitamin K2 according to the forms ethyl ester (EE), triglycerides (TG) and MaxSimil® (monoglycerides, MAG): Calculating the time when the maximum concentration is reached, as the fourth parameter of the PK | Treatments are randomly assigned on days 0, 7 and 14 of the clinical study. GC and HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours post-treatment.
  Plasma Omega-3 (DHA and EPA) will be measured by gas phase chromatography while plasma vitamin K2 will be measured by high-performance liquid chromatography (HPLC), each being performed randomly blindly. After GC and HPLC analyzes, time when the maximum concentration is reached will be calculated, as the fourth parameter of the PK. Statistical analyzes will then be performed on this PK parameter.

SECONDARY OUTCOMES:
To determine the incidence of side effects (including gastrointestinal discomfort) of these same three forms of omega-3 fatty acid supplements | A questionnaire will document the side effects felt by participants during the omega-3 supplement taking day.
  The side effects of EPA + DHA type omega-3 supplements, all mild, belong to the category of gastrointestinal discomfort. These include dysgeusia (fishy taste or taste alteration), belching and nausea. A questionnaire will document the side effects felt by participants during the omega-3 supplement taking day. Statistical analyzes will then be performed on the evaluation of side effects (including gastrointestinal discomfort) by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Plourde, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Melanie Plourde, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data to other researchers

REFERENCES:
- [Derived] Chevalier L, Vachon A, Plourde M. Pharmacokinetics of Supplemental Omega-3 Fatty Acids Esterified in Monoglycerides, Ethyl Esters, or Triglycerides in Adults in a Randomized Crossover Trial. J Nutr. 2021 May 11;151(5):1111-1118. doi: 10.1093/jn/nxaa458. PMID 33564872